CLINICAL TRIAL: NCT01619969
Title: Celgosivir Proof of Concept Trial for Treatment of Acute Dengue Fever
Brief Title: Celgosivir as a Treatment Against Dengue
Acronym: CELADEN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/025/E
Record Dates: First submitted 2012-05-15; First posted 2012-06-15 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — celgosivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celgosivir (Experimental)
  Interventions: Drug: celgosivir
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celgosivir — 100 mg capsules, 400 mg loading dose 200 mg bid
  Other Names: Bu-Cast
  Arms: Celgosivir
Drug: placebo — Capsules of identical appearance containing starch
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Phase 1b Clinical Study to Evaluate the Activity, Pharmacokinetics, Safety and Tolerability of Celgosivir in Adults with Confirmed Dengue Fever.

DETAILED DESCRIPTION:
Patients with confirmed dengue fever who meet all inclusion and exclusion criteria will be enrolled and admitted to the Investigational Medicine Unit. Patients will be randomized 1:1 to celgosivir or placebo. Capsules of placebo or celgosivir will be administered for 5 days. While in hospital, daily clinical exams will be conducted, and blood samples will be collected for viral load, quantitative NS1, hematology, clinical chemistry, cytokine levels and pharmacokinetics (PK). Safety assessments will be conducted. At discharge on Study Day 5, patients will be asked to return on Study Days 7, 10, and 15 for blood sampling and safety assessments.

ELIGIBILITY:
Main Inclusion Criteria:

* Fever of ≥ 38°C of ≤ 48 hr duration.
* At least two of the following criteria indicating probable dengue infection:

  * Live or work in or recent travel to dengue endemic area
  * Nausea and vomiting
  * Presence of rash
  * Aches and pains, including headache, or retro-orbital, muscle or joint pain
* Positive NS1 strip assay

Main Exclusion Criteria:

* Clinical signs and symptoms for severe dengue
* Patients with certain abnormal laboratory values
* History of presently active intestinal disorders
* Severe diarrhea
* Current usage of anticoagulant drugs
* Other clinically significant acute illness
* History of severe drug and/or food allergies
* Exposure to investigational agent within 30 days prior to study drug administration
* Clinically significant abnormal physical exam unrelated to dengue fever
* Pregnancy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Virological Log Reduction (Virological Endpoint) | 4 days
Fever Reduction (Clinical Endpoint) | 4 days

SECONDARY OUTCOMES:
Safety-Proportion of patients experiencing adverse events and serious adverse events | 14 days
  The proportion of patients experiencing adverse events and serious adverse events
Quantitative NS1 and NS1 clearance | 14 days
  NS1 non-structural protein 1
Hematology | 14 days
  Leukocytes, platelets, hematocrit
Pharmacokinetics - Clearance of drug (L/hr) | 5 days
  Clearance of drug (L/hr)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Vasudevan, PhD, Study Director — Duke-NUS Graduate Medical School
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Sung C, Wei Y, Watanabe S, Lee HS, Khoo YM, Fan L, Rathore AP, Chan KW, Choy MM, Kamaraj US, Sessions OM, Aw P, de Sessions PF, Lee B, Connolly JE, Hibberd ML, Vijaykrishna D, Wijaya L, Ooi EE, Low JG, Vasudevan SG. Extended Evaluation of Virological, Immunological and Pharmacokinetic Endpoints of CELADEN: A Randomized, Placebo-Controlled Trial of Celgosivir in Dengue Fever Patients. PLoS Negl Trop Dis. 2016 Aug 10;10(8):e0004851. doi: 10.1371/journal.pntd.0004851. eCollection 2016 Aug. PMID 27509020
- [Derived] Low JG, Sung C, Wijaya L, Wei Y, Rathore APS, Watanabe S, Tan BH, Toh L, Chua LT, Hou Y, Chow A, Howe S, Chan WK, Tan KH, Chung JS, Cherng BP, Lye DC, Tambayah PA, Ng LC, Connolly J, Hibberd ML, Leo YS, Cheung YB, Ooi EE, Vasudevan SG. Efficacy and safety of celgosivir in patients with dengue fever (CELADEN): a phase 1b, randomised, double-blind, placebo-controlled, proof-of-concept trial. Lancet Infect Dis. 2014 Aug;14(8):706-715. doi: 10.1016/S1473-3099(14)70730-3. Epub 2014 May 28. PMID 24877997